CLINICAL TRIAL: NCT02974049
Title: Alternative Chemotherapies for Lymphatic Filariasis (LF) Treatment and Elimination in Africa [Cote d'Ivoire]
Brief Title: Lymphatic Filariasis (LF) in Ivory Coast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Christopher L. King, MD, PhD, Professor of International Health, Medicine and Pathology, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-14-13
Record Dates: First submitted 2016-11-22; First posted 2016-11-28 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2019-04

CONDITIONS: Lymphatic Filariasis
Keywords: Ivermectin; Albendazole; Diethylcarbamazine
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Albendazole; Ivermectin; Diethylcarbamazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Treatment (Active Comparator): Albendazole 400 mg + Ivermectin 200 µg/kg body weight administered annually (at 0, 12 and 24 months)
  Interventions: Drug: Albendazole; Drug: Ivermectin
- ALB 400 mg x2 per year (Experimental): Albendazole 400 mg given at 0, 6, 12, 18, 24 and 30 months
  Interventions: Drug: Albendazole
- ALB 800 mg x2 per year (Experimental): Albendazole 800 mg given at 0, 6, 12, 18, 24 and 30 months
  Interventions: Drug: Albendazole
- ALB 400mg + IVM 200mcg/kg + DEC 6mg/kg (Experimental): Albendazole 400 mg plus Ivermectin 200 µg/kg body weight plus Diethylcarbamazine 6 mg/kg body weight given one time only
  Interventions: Drug: Albendazole; Drug: Ivermectin; Drug: Diethylcarbamazine

INTERVENTIONS:
Drug: Albendazole — Subjects in Arms 1, 2, and 4 will receive 400mg of Albendazole
  Subjects in Arm 3 will receive 800mg of Albendazole
  Other Names: ALB
Drug: Ivermectin — Subjects in Arms 1 and 4 will receive 200mg/kg body weight
  Other Names: IVM
  Arms: ALB 400mg + IVM 200mcg/kg + DEC 6mg/kg; Standard Treatment
Drug: Diethylcarbamazine — Participants in Arm 4 will receive 6mg/kg of Diethylcarbamazine per body weight
  Other Names: DEC
  Arms: ALB 400mg + IVM 200mcg/kg + DEC 6mg/kg

SUMMARY:
The recommended treatment for elimination of LF in sub-Saharan Africa is annual mass drug administration (MDA) with single dose Albendazole (ALB) plus Ivermectin (IVM) given for at least 5-7 years. However, in areas where LF is co-endemic with a related filarial parasite, Loa loa, co-infection with L. loa represents a serious barrier to LF elimination because IVM used in LF MDA can result in severe reactions and even death in individuals with high microfilaria (mf) levels of L. loa. Screening for heavy L. loa infection is problematic. To overcome this problem, monotherapy with ALB is possible, since this drug has little or no effect on circulating mf and thus would not cause adverse effects in people with heavy L. loa infections. Moreover ALB has been shown to have embryostatic or embryocidal effects in female adult worms resulting in decreased mf levels with time as natural attrition of circulating mf occurs. Thus this open-label, randomized clinical trial will examine treatment with ALB monotherapy administered twice per year over a period of 3 years with the primary endpoint being the proportion of individuals with total clearance of mf at 36 months and Alere antigen test negativity (a more sensitive circulating antigen test of filarial infection). Two of the treatment arms will include ALB at two different doses, 400mg or 800mg (fixed dose twice yearly) as compared to standard treatment of ALB (400 mg) plus IVM (150-200 µg/kg) administered annually. Observations from an ongoing clinical trial in Papua New Guinea suggest that a single dose of triple therapy with ALB + IVM + DEC may be highly effective in sterilizing adult female worms. Therefore to confirm and expand these important preliminary observations in a different population, a fourth arm will be included in the current clinical trial in which subjects will receive all three drugs. The clinical trial will be performed in a region of Cote d'Ivoire where onchocerciasis and loiasis are not endemic.

DETAILED DESCRIPTION:
Lymphatic filariasis (LF) is a deforming and disabling infectious disease that causes elephantiasis and genital deformity (especially hydroceles). The infection affects some 120 million people in 81 countries in tropical and subtropical regions with well over 1 billion people at risk of acquiring the disease. LF is caused by Wuchereria bancrofti and Brugia spp. (B. malayi and B. timori), nematode parasites that are transmitted by mosquitoes. The World Health Organization (WHO) developed a plan for LF elimination that is based on using novel approaches to rapidly map endemic areas and 4 to 6 annual rounds of MDA with antifilarial medication. A recent summary from WHO reported that more than 4 billion doses of MDA were distributed between 2000 and 2012. Thus, the Global Program to Eliminate Lymphatic Filariasis (GPELF) is the largest infectious disease intervention program attempted to date based on MDA (Ottesen, Hooper et al.

2008). MDA has worked better in some areas than others. There are a number of challenges faced by GPELF. These include (among others) inability to conduct MDA programs in areas of Africa where L. loa is coendemic because of the unacceptable risk of Serious Adverse Events (SAE's) with IVM in persons with heavy L. loa infections (Hoerauf, Pfarr et al. 2011), the limited macrofilaricidal activity of current MDA regimens (especially ALB + IVM) that necessitate repeated annual rounds of MDA (Geary and Mackenzie , Hoerauf, Pfarr et al. 2011), and the difficulty of achieving high compliance rates for MDA over a period of years (Hoerauf, Pfarr et al. 2011). It is clear that new (or reformulated) drugs and/or dosing schedules for LF MDA have the potential to greatly improve the number of countries that will successfully eliminate LF by the WHO target date of 2020. This is especially important for areas of Central and West Africa where MDA has not been implemented because of the possible co-infection with L. loa and logistical and financial challenges to delivering annual doses of IVM + ALB MDA to millions of individuals over multiple years.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18-70 years
* ≥50 MF/mL based on Nuclepore filtration
* Willing to give informed consent

Exclusion Criteria:

* Prior treatment for LF within last 5 years
* Pregnancy (perform pregnancy test)
* Hemoglobin <7 g/dL
* Permanent disability, serious medical illness that prevents or impedes study participation and/or comprehension
* AST/ALT and creatinine >1.5 upper limit of normal
* Proteinuria or hematuria >3+
* Skin snip positivity for O. volvulus MF

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Total clearance of Microfilariae | 36 months
  The percentage of participants with total clearance of Microfilariae

SECONDARY OUTCOMES:
Total clearance of MF at 24 months | 24 months
  Percentage of subjects with total clearance of MF at 24 months
Percent MF reduction | 24 and 36 months
  Percent MF reduction at 24 and 36 months compared to baseline level
Reduction in W. bancrofti antigen level | 12, 24 and 36 months
  Percent reduction in W. bancrofti antigen level measured by Og4C3 assay at 12, 24 and 36 months compared to baseline level
Alere Filariasis Test Strip negative | 12, 24 and 36 months
  Percentage of subjects that become Alere Filariasis Test Strip negative at 12, 24 and 36 months
reduction in viable worm nests | 12, 24, and 36 months
  Percent reduction in viable worm nests relative to baseline (time 0) based on follow up scrotal ultrasound examination performed at 12, 24 and 36 months
Diversity of parasites | 0 and 36 months
  Diversity of parasites before and after treatment using genetic markers
type and level of parasite-specific host immune response | 0 and 36 months
  Relation of type and level of parasite-specific host immune response with the initial and sustained clearance of parasites

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L King, MD PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Cote d'Ivoire, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
Not personal identifying data but infection levels will be shared.

REFERENCES:
- [Background] Awadzi K, Edwards G, Duke BO, Opoku NO, Attah SK, Addy ET, Ardrey AE, Quartey BT. The co-administration of ivermectin and albendazole--safety, pharmacokinetics and efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2003 Mar;97(2):165-78. doi: 10.1179/000349803235001697. PMID 12803872
- [Background] Awadzi K, Edwards G, Opoku NO, Ardrey AE, Favager S, Addy ET, Attah SK, Yamuah LK, Quartey BT. The safety, tolerability and pharmacokinetics of levamisole alone, levamisole plus ivermectin, and levamisole plus albendazole, and their efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2004 Sep;98(6):595-614. doi: 10.1179/000349804225021370. PMID 15324466
- [Background] Bockarie MJ, Tavul L, Ibam I, Kastens W, Hazlett F, Tisch DJ, Alpers MP, Kazura JW. Efficacy of single-dose diethylcarbamazine compared with diethylcarbamazine combined with albendazole against Wuchereria bancrofti infection in Papua New Guinea. Am J Trop Med Hyg. 2007 Jan;76(1):62-6. PMID 17255231
- [Background] Boussinesq M, Kamgno J, Pion SD, Gardon J. What are the mechanisms associated with post-ivermectin serious adverse events? Trends Parasitol. 2006 Jun;22(6):244-6. doi: 10.1016/j.pt.2006.04.006. Epub 2006 Apr 24. No abstract available. PMID 16632406
- [Background] Chu, B. K., P. J. Hooper, M. H. Bradley, D. A. McFarland and E. A. Ottesen
- [Background] Geary TG. Ivermectin 20 years on: maturation of a wonder drug. Trends Parasitol. 2005 Nov;21(11):530-2. doi: 10.1016/j.pt.2005.08.014. Epub 2005 Aug 26. PMID 16126457
- [Background] Ottesen EA. Lymphatic filariasis: Treatment, control and elimination. Adv Parasitol. 2006;61:395-441. doi: 10.1016/S0065-308X(05)61010-X. PMID 16735170
- [Background] Geary TG, Mackenzie CD. Progress and challenges in the discovery of macrofilaricidal drugs. Expert Rev Anti Infect Ther. 2011 Aug;9(8):681-95. doi: 10.1586/eri.11.76. PMID 21819332
- [Background] Hoerauf A, Pfarr K, Mand S, Debrah AY, Specht S. Filariasis in Africa--treatment challenges and prospects. Clin Microbiol Infect. 2011 Jul;17(7):977-85. doi: 10.1111/j.1469-0691.2011.03586.x. PMID 21722251
- [Background] Hooper PJ, Bradley MH, Biswas G, Ottesen EA. The Global Programme to Eliminate Lymphatic Filariasis: health impact during its first 8 years (2000-2007). Ann Trop Med Parasitol. 2009 Oct;103 Suppl 1:S17-21. doi: 10.1179/000349809X12502035776513. PMID 19843394
- [Background] Horton J. Albendazole: a broad spectrum anthelminthic for treatment of individuals and populations. Curr Opin Infect Dis. 2002 Dec;15(6):599-608. doi: 10.1097/00001432-200212000-00008. PMID 12821837
- [Background] Horton J. The development of albendazole for lymphatic filariasis. Ann Trop Med Parasitol. 2009 Oct;103 Suppl 1:S33-40. doi: 10.1179/000349809X12502035776595. PMID 19843396
- [Background] Hotez PJ, Savioli L, Fenwick A. Neglected tropical diseases of the Middle East and North Africa: review of their prevalence, distribution, and opportunities for control. PLoS Negl Trop Dis. 2012;6(2):e1475. doi: 10.1371/journal.pntd.0001475. Epub 2012 Feb 28. PMID 22389729
- [Background] Kitzman D, Wei SY, Fleckenstein L. Liquid chromatographic assay of ivermectin in human plasma for application to clinical pharmacokinetic studies. J Pharm Biomed Anal. 2006 Mar 3;40(4):1013-20. doi: 10.1016/j.jpba.2005.08.026. Epub 2005 Oct 19. PMID 16242280
- [Background] Mand S, Debrah A, Batsa L, Adjei O, Hoerauf A. Reliable and frequent detection of adult Wuchereria bancrofti in Ghanaian women by ultrasonography. Trop Med Int Health. 2004 Oct;9(10):1111-4. doi: 10.1111/j.1365-3156.2004.01304.x. PMID 15482404
- [Background] McGarry HF, Plant LD, Taylor MJ. Diethylcarbamazine activity against Brugia malayi microfilariae is dependent on inducible nitric-oxide synthase and the cyclooxygenase pathway. Filaria J. 2005 Jun 2;4:4. doi: 10.1186/1475-2883-4-4. PMID 15932636
- [Background] Moreno Y, Nabhan JF, Solomon J, Mackenzie CD, Geary TG. Ivermectin disrupts the function of the excretory-secretory apparatus in microfilariae of Brugia malayi. Proc Natl Acad Sci U S A. 2010 Nov 16;107(46):20120-5. doi: 10.1073/pnas.1011983107. Epub 2010 Nov 1. PMID 21041637
- [Background] Ottesen EA, Duke BO, Karam M, Behbehani K. Strategies and tools for the control/elimination of lymphatic filariasis. Bull World Health Organ. 1997;75(6):491-503. PMID 9509621
- [Background] Ottesen EA, Hooper PJ, Bradley M, Biswas G. The global programme to eliminate lymphatic filariasis: health impact after 8 years. PLoS Negl Trop Dis. 2008 Oct 8;2(10):e317. doi: 10.1371/journal.pntd.0000317. PMID 18841205
- [Background] Teruel M, Dercole J, Catalano R. Evaluation of potential embryo toxicity of albendazole sulphoxide in CF1 mice. Biocell. 2011 Apr;35(1):29-33. PMID 21667669
- [Background] Weil GJ, Curtis KC, Fakoli L, Fischer K, Gankpala L, Lammie PJ, Majewski AC, Pelletreau S, Won KY, Bolay FK, Fischer PU. Laboratory and field evaluation of a new rapid test for detecting Wuchereria bancrofti antigen in human blood. Am J Trop Med Hyg. 2013 Jul;89(1):11-15. doi: 10.4269/ajtmh.13-0089. Epub 2013 May 20. PMID 23690552
- [Background] Zoure HG, Wanji S, Noma M, Amazigo UV, Diggle PJ, Tekle AH, Remme JH. The geographic distribution of Loa loa in Africa: results of large-scale implementation of the Rapid Assessment Procedure for Loiasis (RAPLOA). PLoS Negl Trop Dis. 2011 Jun;5(6):e1210. doi: 10.1371/journal.pntd.0001210. Epub 2011 Jun 28. PMID 21738809
- [Derived] Ouattara AF, Bjerum CM, Aboulaye M, Kouadio O, Marius VK, Andersen B, Lew D, Goss CW, Weil GJ, Koudou BG, King CL. Semiannual Treatment of Albendazole Alone is Efficacious for Treatment of Lymphatic Filariasis: A Randomized Open-label Trial in Cote d'Ivoire. Clin Infect Dis. 2022 Jul 6;74(12):2200-2208. doi: 10.1093/cid/ciab194. PMID 33674871
- [Derived] Bjerum CM, Ouattara AF, Aboulaye M, Kouadio O, Marius VK, Andersen BJ, Weil GJ, Koudou BG, King CL. Efficacy and Safety of a Single Dose of Ivermectin, Diethylcarbamazine, and Albendazole for Treatment of Lymphatic Filariasis in Cote d'Ivoire: An Open-label Randomized Controlled Trial. Clin Infect Dis. 2020 Oct 23;71(7):e68-e75. doi: 10.1093/cid/ciz1050. PMID 31641754